CLINICAL TRIAL: NCT06902103
Title: Pharmacokinetic Study of Single and Multiple Intravenous Administration of Nalbuphine Hydrochloride Injection in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yangtze River Pharmaceutical Group Jiangsu Zilong Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Yangtze River Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: YZJ-NBF-PK-2302
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: Nabufine Hydrochloride Injection
- Group B (Experimental)
  Interventions: Drug: Nabufine Hydrochloride Injection

INTERVENTIONS:
Drug: Nabufine Hydrochloride Injection — PartA: Nabufine Hydrochloride Injection are administered Intravenous injection single dose
  Arms: Group A
Drug: Nabufine Hydrochloride Injection — PartB: Nabufine Hydrochloride Injection are administered Intravenous injection multi dose
  Arms: Group B

SUMMARY:
Objective：To evaluate the pharmacokinetic characteristics and safety of single and multiple intravenous injections of nalbuphine hydrochloride injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 ~ 65 years (inclusive, calculated from the date of signing the informed consent), half males and half females.
2. Weight ≥ 50.0 kg for males, or ≥ 45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 26.0 kg/m2 (inclusive), BMI= weight (kg)/height2(m2).
3. Subjects have no plans to donate sperm or eggs, no plans to become pregnant and voluntarily take effective contraceptive measures (including partners) from signing the informed consent form to 3 months after the last dose of investigational product. See Appendix 2 of the protocol for specific contraceptive measures.
4. Subjects who are able to understand and willing to complete the study in strict compliance with the clinical protocol and sign the informed consent form.

Exclusion Criteria:

1. Subjects with any history of clinically significant diseases or conditions that may affect the test results in the opinion of the investigator, including but not limited to the respiratory system (such as obstructive sleep apnea syndrome, chronic bronchial asthma, etc.), cardiovascular system (such as syncope, etc.), digestive system, endocrine system, nervous system (such as epilepsy), urinary system or blood, immune, mental and metabolic disease history.
2. Subjects with a history of frequent nausea or vomiting of any etiology.
3. Subjects with known history of drug, food or other substance allergy.
4. Subjects who have poor peripheral venous access or have a history of needle and blood fainting.
5. Pregnant or lactating women, or subjects with positive blood pregnancy test results.
6. Subjects with clinically significant abnormal ECG findings at screening, such as QTcF ≥ 450 ms in men, QTcF ≥ 470 ms or PR interval ≥ 200 ms or QRS complex duration ≥ 120 ms in women.
7. Subjects with abnormal vital signs at screening (systolic blood pressure < 90 mmHg or > 140 mmHg, diastolic blood pressure < 50 mmHg or > 90 mmHg; pulse < 50 beats/min or > 100 beats/min) or physical examination, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function), chest anteroposterior abnormal subjects with clinical significance (based on the judgment of clinicians).
8. Those who are positive in any index screening of hepatitis B virus surface antigen, Treponema pallidum-specific antibody, human immunodeficiency virus antibody, or hepatitis C virus antibody at screening.
9. Subjects with positive urine drug screening or any history of drug abuse within 1 year prior to screening.
10. Subjects who frequently consume alcohol within 6 months prior to screening, i.e., consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% spirits, alcohol or 150 mL of wine), or whose alcohol breath test result > 0.0 mg/100 mL, or take any alcohol-containing products within 48 hours before the first use of investigational products, or who cannot stop using any alcohol products during the study.
11. Subjects smoke an average of 5 or more cigarettes per day within 3 months prior to screening, or who have used tobacco products within 48 hours before the first use of investigational products, or those who cannot stop using any tobacco products during the study.
12. Subjects who have donated blood or experienced massive blood loss (> 400 mL, excluding blood loss during menstruation in women), received blood transfusions or used blood products within 3 months prior to screening.
13. Subjects who participated in any clinical trial and administered investigational drugs or investigational medical devices within 3 months prior to screening.
14. Subjects who have undergone surgical procedures within 4 weeks prior to screening, or plan to undergo surgical procedures during the study period.
15. Subjects who have received attenuated/DNA nucleic acid/recombinant protein vaccination within 4 weeks before screening, or inactivated vaccination within 2 weeks before screening, or plan to receive any vaccination during the study period.
16. Subjects who have taken any drugs that inhibit or induce CYP or UGT enzymes within 28 days prior to screening.
17. Subjects who have taken any prescription drugs, over-the-counter drugs, health products, vitamins, and Chinese herbal medicines within 14 days before the first use of investigational product.
18. Subjects who have consumed grapefruit, pomelo, pitaya, mango and other fruits or related products affecting metabolic enzymes within 7 days before the first use of investigational products。
19. Subjects who have taken any food or beverage rich in caffeine or xanthine (coffee, tea, cola, chocolate, etc.) within 48 hours before the first use of investigational product, or who do not agree to avoid eating the above food or beverage during the trial.
20. Subjects who are not suitable for participating in this clinical trial in the investigator 's opinion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum drug plasma concentration) | up to 12 hours after first administration
AUC0-t (Total area under the plasma drug concentration-time curve from time of administration to the time of the last quantifiable drug concentration) | up to 12 hours after first administration
AUC0-∞ (Total area under the plasma drug concentration-time curve) | up to 12 hours after first administration
Tmax (Time to achieve Cmax) | up to 12 hours after first administration
T1/2z (Apparent terminal elimination half-life) | up to 12 hours after first administration
AUC_%Extrap (The percentage of the portion estimated through extrapolation) | up to 12 hours after first administration
MRT (Mean residence time) | up to 12 hours after first administration
CLz (Clearance of the analyte in plasma) | up to 12 hours after first administration
Occurence of adverse events | up to 5 days for part A, up to 7 days for part B

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, China